CLINICAL TRIAL: NCT05154955
Title: A Multi-Center, Randomized, Double-Blinded, Vehicle-Controlled Study of the Safety and Efficacy of 10XB-101 in Adult Subjects With Submental Fat
Brief Title: A Safety and Tolerability Study of 10XB-101 Injection in Adult Subjects With Submental Fat
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 10xBio, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 210-9451-203
Record Dates: First submitted 2021-12-01; First posted 2021-12-13 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-06

CONDITIONS: Submental Fat
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 10XB-101 Solution for Injection, 2.0% (Experimental): Participants receive 10XB-101 Solution for Injection, 2.0% via subcutaneous injection up to 10 mL. Injection treatment will occur once every 4-6 weeks for up to 6 treatments.
  Interventions: Drug: 10XB-101 Solution for Injection
- 10XB-101 Solution for Injection, 3.0% (Experimental): Participants receive 10XB-101 Solution for Injection, 3.0% via subcutaneous injection up to 10 mL. Injection treatment will occur once every 4-6 weeks for up to 6 treatments.
  Interventions: Drug: 10XB-101 Solution for Injection
- 10XB-101 Solution for Injection, 4.5% (Experimental): Participants receive 10XB-101 Solution for Injection, 4.5% via subcutaneous injection up to 10 mL. Injection treatment will occur once every 4-6 weeks for up to 6 treatments.
  Interventions: Drug: 10XB-101 Solution for Injection
- 10XB-101 Vehicle Solution for Injection (Placebo Comparator): Participants receive 10XB-101 Vehicle Solution for Injection, via subcutaneous injection up to 10 mL. Injection treatment will occur once every 4-6 weeks for up to 6 treatments.
  Interventions: Drug: 10XB-101 Vehicle Solution for Injection

INTERVENTIONS:
Drug: 10XB-101 Solution for Injection — One of the three concentrations of 10XB-101 will be evaluated against placebo for submental fat reduction.
  Arms: 10XB-101 Solution for Injection, 2.0%; 10XB-101 Solution for Injection, 3.0%; 10XB-101 Solution for Injection, 4.5%
Drug: 10XB-101 Vehicle Solution for Injection — This is the placebo control
  Arms: 10XB-101 Vehicle Solution for Injection

SUMMARY:
The purpose of this research study is to determine the safety and efficacy of 10XB-101 vs. vehicle (placebo) for adults with excessive submental fat (SMF).

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or non-pregnant female 18 to 65 years old.
* Subject has provided written informed consent.
* Subject has qualifying Submental Fat evaluation score.
* Subject has had a stable body weight for the past 6 months prior to starting study.
* Subject is willing to undergo test article injections as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.

Exclusion Criteria:

* Subject is pregnant, lactating, or is planning to become pregnant during the study.
* Subject has loose skin in the submental area, diffuse SMF, or prominent platysmal bands at rest that may interfere with evaluation of localized fat, in the opinion of the investigator.
* Subject has had any prior treatment for SMF (e.g., deoxycholic acid, cryotherapy, liposuction, surgery).
* Subject has any medical condition that affects clotting and/or platelet function
* Subject has a history of allergy or sensitivity to polidocanol or any of the other ingredients in the test articles.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Clinician Submental Fat Scale (CSFS) | 24 weeks after final injection treatment
  Change from Baseline after final treatment. CSFS is a 5 point scale, with a higher score indicating higher severity
Patient Submental Fat Scale (PSFS) | 24 weeks after final injection treatment
  Change from Baseline after final treatment. PSFS is a 5 point scale, with a higher score indicating higher severity

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Site 03, Encino, California
  - Site 02, San Diego, California
  - Site 01, San Diego, California
  - Site 04, Rolling Meadows, Illinois

IPD SHARING:
Plan to Share IPD: No